CLINICAL TRIAL: NCT01219504
Title: Evaluation of the Impact of Embryo Biopsy on the Reproductive Potential of Embryos Undergoing IVF
Brief Title: Evaluation of the Impact of Embryo Biopsy on the Reproductive Potential of Embryos Undergoing In Vitro Fertilization (IVF)
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-17
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Each Patient is Both Case and Control; 1 Embryo Will be Biopsied and 1 Embryo is Not
Keywords: PGD; IVF

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples on female and male patients. Buccal swabs on infant(s).
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the impact of embryo biopsy on the reproductive potential of human embryos.

DETAILED DESCRIPTION:
This study will recruit patients from the NY/NJ/CT/eastern PA area only.

All patients will undergo an in vitro fertilization (IVF) cycle with hormonal stimulation and an egg retrieval procedure as deemed appropriate for their diagnosis. Following biopsy, the embryos will be transferred. There will be no delay in the time of transfer as no cells will be analyzed prior to transfer.

On day 3 or day 5 of embryo development, all patients will undergo a two (2) embryo transfer. The embryos selected for transfer will be the 2 morphologically best of the embryo cohort. Once selected for transfer, the embryos will be randomized so that one will be biopsied and the other will be transferred without undergoing biopsy. The embryo randomized to biopsy will have a single cell biopsied.

Following delivery, buccal swabs will be collected from infants.

ELIGIBILITY:
This study will recruit patients from the NY/NJ/CT/eastern PA area only.

Inclusion Criteria:

1. Maximum of one prior failed IVF treatment cycle
2. Female partner less than 35 years of age
3. Normal day 3 FSH level (<10 miu/mL)
4. Total basal antral follicle count greater than or equal to 12
5. Male partner with greater than 100,000 total motile spermatozoa and at least 1% normal forms
6. Body mass index (BMI) < or = 32
7. Normal uterine cavity

Exclusion Criteria:

1. Diagnosis of chronic anovulation secondary to polycystic ovarian disease
2. Diagnosis of endometrial insufficiency
3. Clinical indication for pre-implantation genetic diagnosis (PGD) (undergoing IVF with PGD to rule out a known genetic defect)
4. Use of testicular aspiration or biopsy procedures to obtain sperm

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 200 infertile couples undergoing IVF will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Impact of biopsy on pregnancy | 1 year
  Impact of the biopsy of the embryo on whether a pregnancy is obtained
Impact of biopsy on delivery | 1 year
  Impact of the biopsy on pregnancy resulting in delivery

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (3):
- United States (3):
  - Reproductive Medicine Associates of Connecticut, Norfolk, Connecticut
  - Reproductive Medicine Associates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associates of New York, New York, New Jersey

REFERENCES:
- [Derived] Scott RT Jr, Upham KM, Forman EJ, Zhao T, Treff NR. Cleavage-stage biopsy significantly impairs human embryonic implantation potential while blastocyst biopsy does not: a randomized and paired clinical trial. Fertil Steril. 2013 Sep;100(3):624-30. doi: 10.1016/j.fertnstert.2013.04.039. Epub 2013 Jun 15. PMID 23773313